CLINICAL TRIAL: NCT01454557
Title: The Effect of Auditory Stimuli on Heart Rate Variability (HRV) During Resting and During Physical Activity Among Patients With Acquired Brain Injury (ABI)
Brief Title: The Effect of Auditory Stimuli on Heart Rate Variability (HRV) Among Patients With Acquired Brain Injury (ABI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ofer Keren, The head of the TBI rehabilitation department, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-11-8846-OK-CTIL
Record Dates: First submitted 2011-10-10; First posted 2011-10-19 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Acquired Brain Injury
Keywords: Acquired Brain Injury; Heart Rate Variability (HRV); Auditory Stimuli; Physical Activity
MeSH Terms: conditions — Brain Injuries; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acquired Brain Injury (Experimental): auditory stimuli for ABI group
  Interventions: Other: Auditory Stimuli
- Controls (Experimental): Auditory stimuli for control group
  Interventions: Other: Auditory Stimuli

INTERVENTIONS:
Other: Auditory Stimuli — Auditory Stimuli during rest and during physical activity

SUMMARY:
Heart Rate Variability (HRV) reflects the responsiveness of the autonomic system to an external stimuli. The aim of this system is to maintain homeostasis.The variability implies on the interaction between the sympathetic and the parasympathetic systems to maintain the ongoing changes of the autonomic system. Following Acquired Brain Injury (ABI), there can be a damage to the Central Nervous System (CNS) function. The damages described in the literature are cognitive, motor and behavioural function, while there is less relation to the autonomic system. The autonomic system can influence the ability of patient with ABI to participate in the rehabilitation program. The aim of this work is to investigate the activity of the autonomic system activity as manifested by HRV among patients with ABI in different conditions: resting, during activity and while listening to different auditory stimuli.

ELIGIBILITY:
Inclusion Criteria:

* 2-4 months from acceptance to rehabilitation medical stable

Exclusion Criteria:

* medical unstable a significant hearing deficit premorbid neurological or mental condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | first measurement: 2 weeks to 2 months from hospitalization to the department: 24 hours EKG follow up for HRV base line. Last measurement: before the release from rehabilitation (up to 12 months).
  Heart Rate Variability as measured by HOLTER EKG during the 4 different conditions: first measuerement 2-8 weeks from hospitalization in the TBI rehabilitation department-24 hours detection for HRV baseline. Second measurement: a week after: EKG during the 4 conditions. Third measurement:a month after the first measure, Fourth measurement: 2 months after the first one. Last measurement: Before the release home from rehabilitation (up to one year from the first measurement).

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Keren, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel